CLINICAL TRIAL: NCT04825054
Title: Cardiopulmonary Effect of Mechanical Ventilation in Children Underwent Surgical Repair of Right Ventricular Hypertrophy: Compared With Pressure Control Ventilation, Pressure Support Ventilation and Neurally Adjusted Ventilatory Assist
Brief Title: Cardiopulmonary Effect of Mechanical Ventilation in Children With Right Ventricular Hypertrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Limin Zhu (Other)
Responsible Party: Sponsor-Investigator, Limin Zhu, Deputy chief physician, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: SCMC-CHC2021006
Record Dates: First submitted 2021-03-01; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Heart-lung Interaction; Right Ventricular Hypertrophy; Postoperative Care; Congenital Heart Disease; Mechanical Ventilation
MeSH Terms: conditions — Hypertrophy, Right Ventricular; Heart Defects, Congenital | interventions — Respiration, Artificial

STUDY DESIGN:
Intervention Model Description: 1. pressure control ventilation
  2. pressure support ventilation
  3. neurally adjusted ventilatory assist
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A 60-min trial ventilated with NAVA (Experimental): Patients underwent surgical repair of right ventricular hypertrophic congenital heart disease. Each patient will undergo three 60-min trials with 30-min wash out during the study period in randomized order. The cardiac output and volume status will be evaluated by a transpulmonary thermodilution device through a pulse contour cardiac output (PiCCO) catheter at the last 10min of each trial. At the mean while an arterial blood gas and echocardiography will perform.
  Interventions: Device: Mechanical ventilation with NAVA mode
- A 60-min trial ventilated with PCV (Experimental): Patients underwent surgical repair of right ventricular hypertrophic congenital heart disease. Each patient will undergo three 60-min trials with 30-min wash out during the study period in randomized order. The cardiac output and volume status will be evaluated by a transpulmonary thermodilution device through a pulse contour cardiac output (PiCCO) catheter at the last 10min of each trial. At the mean while an arterial blood gas and echocardiography will perform.
  Interventions: Device: Mechanical ventilation with PCV mode
- A 60-min trial ventilated with PSV (Experimental): Patients underwent surgical repair of right ventricular hypertrophic congenital heart disease. Each patient will undergo three 60-min trials with 30-min wash out during the study period in randomized order. The cardiac output and volume status will be evaluated by a transpulmonary thermodilution device through a pulse contour cardiac output (PiCCO) catheter at the last 10min of each trial. At the mean while an arterial blood gas and echocardiography will perform.
  Interventions: Device: Mechanical ventilation with PSV mode

INTERVENTIONS:
Device: Mechanical ventilation with NAVA mode — To compare the hemodynamic and pulmonary effect in patients after surgical repair with right ventricular hypertrophic ventilated with PCV, PSV and NAVA by a crossover study.
  Each patient will undergo three 60-min trials during the study period in randomized order. The cardiac output and volume status will be evaluated by a transpulmonary thermodilution device through a pulse contour cardiac output (PiCCO) catheter at the last 10min of each trial. At the mean while an arterial blood gas and echocardiography will perform.
  Arms: A 60-min trial ventilated with NAVA
Device: Mechanical ventilation with PCV mode — To compare the hemodynamic and pulmonary effect in patients after surgical repair with right ventricular hypertrophic ventilated with PCV, PSV and NAVA by a crossover study.
  Each patient will undergo three 60-min trials during the study period in randomized order. The cardiac output and volume status will be evaluated by a transpulmonary thermodilution device through a pulse contour cardiac output (PiCCO) catheter at the last 10min of each trial. At the mean while an arterial blood gas and echocardiography will perform.
  Arms: A 60-min trial ventilated with PCV
Device: Mechanical ventilation with PSV mode — To compare the hemodynamic and pulmonary effect in patients after surgical repair with right ventricular hypertrophic ventilated with PCV, PSV and NAVA by a crossover study.
  Each patient will undergo three 60-min trials during the study period in randomized order. The cardiac output and volume status will be evaluated by a transpulmonary thermodilution device through a pulse contour cardiac output (PiCCO) catheter at the last 10min of each trial. At the mean while an arterial blood gas and echocardiography will perform.
  Arms: A 60-min trial ventilated with PSV

SUMMARY:
Neurally adjusted ventilatory assist (NAVA) is a new mode of mechanical ventilation that delivers ventilatory assist in proportion to neural effort. The investigators hope to compare the hemodynamic and pulmonary effect in children after surgical repair of congenital heart disease with right ventricular hypertrophic ventilated with Pressure control ventilation (PCV), Pressure support ventilation (PSV), and NAVA by a crossover study.

DETAILED DESCRIPTION:
In the patients suffered from congenital heart disease with right ventricular hypertrophy, the preload of the heart will be influenced by the variation of the intrathoracic pressure. The cardiopulmonary interaction during mechanical ventilation will be an important influence factor on hemodynamics after surgical repair for these patients. As a new mode of mechanical ventilation, NAVA delivers ventilatory assist in proportion to patients' neural effort avoiding over ventilation.

The investigators designed a crossover study to evaluate the cardiopulmonary effect in patients with congenital heart disease with right ventricular hypertrophy when ventilated with NAVA postoperatively, compared with the conventional mode of pressure control ventilation and pressure support ventilation. Each patient will undergo three 60-min trials during the study period in randomized order. The cardiac output and volume status will be evaluated by a transpulmonary thermodilution device through a pulse contour cardiac output (PiCCO) catheter at the last 10min of each trial. At the mean while an arterial blood gas and echocardiography will perform.

Data are expressed as mean ± standard deviation. Datas from the three registrations will be compared using a repeated-measures ANOVA. The comparison of each mode will be assessed by the SNK methods post hoc test. A p value of less than 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients underwent surgical repair of right ventricular hypertrophic congenital heart disease
2. Obtain informed consent signed by parents

Exclusion Criteria:

1. Significant residual shunt (more than 2mm), residual obstruction of right ventricular outflow tract (RVOT) or A-V valve insufficiency.
2. Hemodynamic instability (whose inotropic score more than 20);
3. Significant bleed (whose chest drainage more than 5ml/kg/h);
4. Failed to insert the PiCCO catheter
5. Dysfunction and abnormal of esophage;
6. Inclusion in other research protocol

Ages: 3 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac output index | Within 72 hours after opeartion
  Cardiac output index messured by PiCCO and echocariography should be improved when ventilated with NAVA or PSV compared with PCV.

SECONDARY OUTCOMES:
Peak inspiratory pressure | Within 72 hours after opeartion
  Peak inspiratory pressure (PIP) should be recorded at the last 3 minutes ventilated with NAVA, PCV or PSV. The average of PIP and MAP of every breath within 3 min will be regarded as the airway pressure of every trial. Data are expressed as mean ± standard deviation. Datas from the three registrations will be compared using a repeated-measures ANOVA. The comparison of each mode will be assessed by the SNK methods post hoc test. A p value of less than 0.05 was considered significant.
Mean airway pressure | Within 72 hours after opeartion
  Mean Airway pressure (MAP) should be recorded at the last 3 minutes ventilated with NAVA, PCV or PSV. The average of PIP and MAP of every breath within 3 min will be regarded as the airway pressure of every trial. Data are expressed as mean ± standard deviation. Datas from the three registrations will be compared using a repeated-measures ANOVA. The comparison of each mode will be assessed by the SNK methods post hoc test. A p value of less than 0.05 was considered significant.
Arterial partial pressure of oxygen | Within 72 hours after opeartion
  The arterial blood gas will be sampled at the last 5 min of every trial. Arterial partial pressure of oxygen (PaO2) of the blood gas analysis during different ventilatory mode of NAVA, PCV or PSV will be compared. Data are expressed as mean ± standard deviation. Datas from the three registrations will be compared using a repeated-measures ANOVA. The comparison of each mode will be assessed by the SNK methods post hoc test. A p value of less than 0.05 was considered significant.
Arterial partial pressure of carbon dioxide | Within 72 hours after opeartion
  The arterial blood gas will be sampled at the last 5 min of every trial. Arterial partial pressure of carbon dioxide (PaCO2) of the blood gas analysis during different ventilatory mode of NAVA, PCV or PSV will be compared. Data are expressed as mean ± standard deviation. Datas from the three registrations will be compared using a repeated-measures ANOVA. The comparison of each mode will be assessed by the SNK methods post hoc test. A p value of less than 0.05 was considered significant.
Arterial oxygen saturation | Within 72 hours after opeartion
  The arterial blood gas will be sampled at the last 5 min of every trial. Arterial oxygen saturation (SaO2) of the blood gas analysis during different ventilatory mode of NAVA, PCV or PSV will be compared. Data are expressed as mean ± standard deviation. Datas from the three registrations will be compared using a repeated-measures ANOVA. The comparison of each mode will be assessed by the SNK methods post hoc test. A p value of less than 0.05 was considered significant.
Lactate | Within 72 hours after opeartion
  The datas of organ purfusion such as lactate during different ventilatory mode of NAVA, PCV or PSV will be gathered from the blood sample at the last 5 min of every trial. Datas from the three registrations will be compared using a repeated-measures ANOVA. The comparison of each mode will be assessed by the SNK methods post hoc test. A p value of less than 0.05 was considered significant.
ScvO2 | Within 72 hours after opeartion
  The datas of organ purfusion such as ScvO2 during different ventilatory mode of NAVA, PCV or PSV will be gathered from the blood sample at the last 5 min of every trial. Datas from the three registrations will be compared using a repeated-measures ANOVA. The comparison of each mode will be assessed by the SNK methods post hoc test. A p value of less than 0.05 was considered significant.
Urine output | Within 72 hours after opeartion
  The total urine output during different ventilatory mode of NAVA, PCV or PSV will be recorded. Datas from the three registrations will be compared using a repeated-measures ANOVA. The comparison of each mode will be assessed by the SNK methods post hoc test. A p value of less than 0.05 was considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Limin Zhu, M.D., Study Director — Shanghai Children/s Medical Center, Shanghai Jiaotong University School of Medicine; Xiaolei Gong, M.D., Principal Investigator — Shanghai Children/s Medical Center, Shanghai Jiaotong University School of Medicine; Zhuoming Xu, Ph. D & M.D., Study Chair — Shanghai Children/s Medical Center, Shanghai Jiaotong University School of Medicine
Locations (2):
- China (2):
  - Cardiac intensive care unit, Department of cardiothoracic vascular surgery, Shanghai Children's Medical Center, Medical college of Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai Children's Medical Center, Shanghai Jiaotong Universiry School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gong X, Zhu L, Zhang M, Liu Y, Li C, Xu Z, Zheng J. Utilizing Spontaneous Ventilation Modes in Patients Underwent Corrective Surgery for Right Ventricular Outflow Tract Obstructive Congenital Heart Disease: A Crossover Study. Rev Cardiovasc Med. 2023 May 11;24(5):143. doi: 10.31083/j.rcm2405143. eCollection 2023 May. PMID 39076742